CLINICAL TRIAL: NCT04744181
Title: Patient Blood Management In CARdiac sUrgical patientS: the ICARUS Study
Brief Title: Patient Blood Management In CARdiac sUrgical patientS
Acronym: ICARUS
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CORSI FILIPPO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0047459/20
Record Dates: First submitted 2021-01-31; First posted 2021-02-08 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Anemia; Blood Loss Anemia; Iron-deficiency; Iron Deficiency Anemia; Iron Deficiency Anemia Treatment; Erythropoiesis Abnormal
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Vitamin B Complex; Folic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cases: patients who fulfill the inclusion criteria
  Interventions: Drug: Ferric carboxymaltose; Drug: B vitamin; Drug: Folic acid
- controls: Patients who underwent cardiac surgery in 2019 and 2018, with an unknown iron status and never treated with iron supplementation.

INTERVENTIONS:
Drug: Ferric carboxymaltose — administration of a single dose of ferric carboxymaltose in those patietns who fulfill the inclusion criteria
  Other Names: ferinject
  Groups: cases
Drug: B vitamin — administration of a single dose of B vitamin in those patietns who fulfill the inclusion criteria
  Groups: cases
Drug: Folic acid — administration of a single dose of folic acid in those patietns who fulfill the inclusion criteria
  Groups: cases

SUMMARY:
Nowadays up to 40% of patients undergoing cardiac surgery receives at least 1 unit of red blood cell transfusion during surgery or during the first week after surgery. Moreover up to 40% of these patients shows an absolute or relative iron deficiency, with or without anaemia.

The objective of this study is to assess whether to implement an adequate correction of iron according to current "patients blood management" recommendations might reduce RBC transfusion requirements in patients undergoing heart surgery.

Data obtained in patients included in the study will be compared to those of a case-control population selected from patients consecutively treated at the same department in the previous 2 years.

DETAILED DESCRIPTION:
Anemia is defined by the World Health Organization (WHO) as a value of hemoglobin (Hb) < 130 g/L in men and < 120 g/L in women. Anemia in surgical patients is a common and serious problem, in fact up to 40% of patients presenting for major surgery are anemic. Patients with pre-operative anemia have significantly higher rates of morbidity and mortality and are likely to receive red blood cell (RBC) transfusions. In turn, RBC are independently associated with worse outcome. Preoperative anemia mainly results from inadequate erythropoiesis owing to iron deficiency. Iron deficiency anemia (IDA) has a complex origin, including either absolute or functional iron deficiency (or iron sequestration). In absolute iron deficiency, iron stores are severely decreased, resulting in anaemia (IDA). Conversely, functional iron deficiency refers to insufficient iron mobilization despite normal or elevated iron stores (iron deficient erythropoiesis, IDE).The most rapid and simple method to correct anaemia is RBC transfusion. More than 30% of cardiac patients receives blood products in the peri-operative phase. However, blood transfusion itself is not without risk: in the setting of cardiac patients, even a single unit of blood transfused is reported to be associated to increased morbidity and mortality. Specifically, blood transfusions in cardiac surgery are associated with infections, ischemic postoperative morbidity, hospital stay, increased early and late mortality, and greater hospital costs. Preoperative correction of iron deficiency, with or without anaemia, is an integral part of the concept of the Patient Blood Management (PBM). Iron supplementation would increase the availability of iron stores and would trigger the process of erythropoiesis; the consequent relative lack of vitamin B12 and folic acid makes fundamental to restore also these 2 vitamins.

The objective of this study is to assess whether to implement an adequate correction of IDA and IDE according to current PBM recommendations might reduce RBC transfusion requirements in patients undergoing heart surgery. Data obtained in patients included in the study will be compared to those of a case-control population selected from patients consecutively treated at the same department in the previous 2 years.

ELIGIBILITY:
Inclusion Criteria:

- all adult patients candidate to planned heart surgery

Exclusion Criteria:

* Pregnancy
* Know allergy to iron, or B vitamin, or folic acid
* Hyperferritinemia (ferritin blood value > 300 ng/ml).
* patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients candidate to planned heart surgery in our tertiary care hospital are eligible for the study purpose.
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving RBC transfusion within post-operative day 7 | within post operative day 7
  Percentage of patients receiving RBC transfusion within post-operative day 7

SECONDARY OUTCOMES:
Hb values at last postoperative control within 7 days from surgery | within post operative day 7
  Hb values at last postoperative control within 7 days from surgery
length of stay in ICU | through study completion, an average of 1 year
  length of stay in ICU
number of allogeneic blood products administered | within the first 7 days post operative
  number of allogeneic blood products administered
duration of mechanical ventilation | within the first 7 days post operative
  duration of mechanical ventilation
acute kidney injury | within the first 7 days post operative
  worsening of renal function
serious adverse events | within the first 12 hours after administration
  including hypersensitivity reactions
infections requiring antibiotic treatment | within the first 7 days post operative
  infections requiring antibiotic treatment
mortality | within the first 7 days after surgery
  patients died within the first 7 days after surgery
major adverse cardiac and cerebrovascular events | within the first 7 days after surgery
  cardiogenic shock, neurological events
cost for the IDA/IDE treatment and blood product costs | within the first 7 days after surgery
  cost for the IDA/IDE treatment and blood product costs

CONTACTS AND LOCATIONS:
Overall Officials: filippo corsi, Dr, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- FPG Fondazione Policlinico Gemelli IRCCS, Roma, roma, Italy

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon reasonable request to the PI and after approval by ethic committee.

REFERENCES:
- [Background] Spahn DR, Schoenrath F, Spahn GH, Seifert B, Stein P, Theusinger OM, Kaserer A, Hegemann I, Hofmann A, Maisano F, Falk V. Effect of ultra-short-term treatment of patients with iron deficiency or anaemia undergoing cardiac surgery: a prospective randomised trial. Lancet. 2019 Jun 1;393(10187):2201-2212. doi: 10.1016/S0140-6736(18)32555-8. Epub 2019 Apr 26. PMID 31036337
- [Derived] Corsi F, Pasquini A, Guerrera M, Bevilacqua F, Taccheri T, Antoniucci ME, Calabrese M, Valentini CG, Orlando N, Bartolo M, Cannetti G, Pellegrino C, Cavaliere F, Teofili L. Single shot of intravenous iron in cardiac surgery: The ICARUS study. J Clin Anesth. 2023 Feb;84:111009. doi: 10.1016/j.jclinane.2022.111009. Epub 2022 Nov 16. PMID 36401886
- See also: Haemoglobin concentration for the diagnosis of anaemia and assesment of severity — https://apps.who.int/iris/bitstream/handle/10665/85839/WHO_NMH_NHD_MNM_11.1_eng.pdf?ua=1
- See also: Perioperative Anemia Management as Part of PBM in Cardiac Surgery - A Narrative Updated Review — https://linkinghub.elsevier.com/retrieve/pii/S1053-0770(19)30639-1
- See also: The impact of anaemia and intravenous iron replacement therapy on outcomes in cardiac surgery — https://research-repository.uwa.edu.au/en/publications/the-impact-of-anaemia-and-intravenous-iron-replacement-therapy-on
- See also: Does the severity of preoperative anemia or blood transfusion have a stronger impact on long-term survival after cardiac surgery? — https://linkinghub.elsevier.com/retrieve/pii/S0022-5223(16)30564-5
- See also: Impact of Preoperative Iron Deficiency on Blood Transfusion in Elective Cardiac Surgery — https://linkinghub.elsevier.com/retrieve/pii/S1053-0770(19)30108-9
- See also: Iron deficiency impairs contractility of human cardiomyocytes through decreased mitochondrial function — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5993224/
- See also: Liberal transfusion strategy to prevent mortality and anaemia-associated, ischaemic events in elderly non-cardiac surgical patients - the study design of the LIBERAL-Trial — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-019-3200-3
- Available data/document: Individual Participant Data Set — https://redcap-irccs.policlinicogemelli.it/